CLINICAL TRIAL: NCT06823622
Title: Evaluation of the Digital Delivery of Person-centered Transitional Care to Empower Adolescents With Chronic Childhood-onset Diseases: The Digi-STEPSTONES Study
Brief Title: Digital Delivery of Person-centered Transitional Care
Acronym: DigiStep
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Digi Stepstones
Record Dates: First submitted 2024-09-12; First posted 2025-02-12 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Asthma in Children; Transplantation
Keywords: Transition; Transfer; Chronic condition; Adolescents; Youth; Young people; Transition program
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Intervention Model Description: A two-arm, comparative, non-inferiority study, using a causal inference methodology will be performed. Arm A involves a pre-test/post-test design where individuals will participate in the digital delivery of the transition program. Arm B is a historical comparison cohort that includes participants from two previous RCTs who received the intervention (the transition program) in-person.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Arm A involves a pre-test/post-test design where individuals will participate in the digital delivery of the transition program.
  Interventions: Behavioral: Stepstones transition program
- Arm B (Other): Arm B is a historical comparison cohort that includes participants from two previous RCTs who received the intervention (the transition program) in-person.
  Interventions: Behavioral: Stepstones transition program

INTERVENTIONS:
Behavioral: Stepstones transition program — The STEPSTONES transition program is an 8-component intervention designed to support adolescents with chronic conditions transitioning to adult care. It includes: a transition coordinator (TC), education about the condition, phone support, guidance on transitioning to adult care, parental guidance, peer meetings, a personalized transition plan, and the actual transfer to adult care. The intervention is implemented in five steps, starting with outpatient visits and culminating in the transfer to adult care. Delivered via the "Mitt vårdmöte" digital platform, the program includes the HEADDDSS adolescent health interview and is conducted by trained specialized nurses.

SUMMARY:
Advances in medical care have extended the life expectancy of individuals with congenital and pediatric-onset diseases, leading to an increased need for effective transition programs as these individuals move from pediatric to adult healthcare. The STEPSTONES project in Sweden is designed to evaluate the effectiveness of a person-centered transition program to support teenagers with chronic conditions during this transition. The project's innovative digital adaptation, Digi-STEPSTONES, seeks to address challenges related to accessibility and continuity of care by delivering the program remotely. This study will assess the non-inferiority of the digital program compared to traditional, in-person care, focusing on outcomes such as patient empowerment, transition readiness, and quality of life. Additionally, the project will explore the implementation and scalability of the digital transition model across various chronic conditions. Preliminary studies have highlighted the importance of structured, person-centered care in improving empowerment and other outcomes in adolescents with chronic illnesses. The Digi-STEPSTONES project aims to provide crucial evidence for the digital delivery of transition programs, potentially enhancing the accessibility and effectiveness of care for young people with chronic conditions in Sweden.

DETAILED DESCRIPTION:
Medical and surgical advances have significantly increased the life expectancy of individuals with congenital and pediatric-onset diseases, often resulting in chronic conditions. Effective lifetime care is crucial, especially during the transition from pediatric to adult care. Transition is a process where adolescents with chronic conditions are prepared to manage their health and life as they move to adult healthcare environments. Transition programs are designed to assist in this preparation, and over the past decade, several randomized-controlled trials (RCTs) have demonstrated the effectiveness of such programs in improving outcomes like self-management, knowledge of the condition, clinic attendance, and satisfaction with care.

In Sweden, the STEPSTONES (Swedish Transition Effects Project Supporting Teenagers with chrONic mEdical conditionS) project is evaluating a person-centered transition program tailored for young individuals with chronic conditions. The project has focused on conditions like congenital heart disease and type 1 diabetes through RCTs and is now exploring a digital adaptation called Digi-STEPSTONES, which aims to deliver the transition program remotely to improve accessibility and continuity of care.

PURPOSE AND AIMS

The main goal of this project is to evaluate the effectiveness of a digitally delivered, person-centered transition program for adolescents with asthma/allergy and those who have undergone a solid organ transplant in a real-world setting. The specific objectives are:

* To investigate the non-inferiority of the digital delivery compared to in-person delivery.
* To evaluate the implementation process of the digital transition program.

SIGNIFICANCE AND NOVELTY Digi-STEPSTONES aligns with person-centered care principles by supporting shared decision-making and empowering adolescents to actively participate in their healthcare. This project is novel as it is the first to provide evidence on the effectiveness of a digitally delivered person-centered transition program, covering multiple conditions, which enhances the generalizability of the findings.

RESEARCH DESIGN AND METHODS

To achieve the project's objectives, two studies will be conducted:

Study 1: Comparative Effectiveness Research (Non-Inferiority Trial) A two-arm, non-inferiority study using a causal inference methodology will be performed. Arm A involves a digital delivery of the transition program, while Arm B is a historical cohort from previous RCTs that received in-person delivery.

The STEPSTONES transition program includes eight components implemented in five steps, and the intervention will be delivered via the "Mitt vårdmöte" platform, already in use for digital healthcare appointments in Sweden. Assessments will be made at ages 16 and 18.5, focusing on primary outcomes like patient empowerment and secondary outcomes like transition readiness, quality of life, and health literacy.

Study 2: Evaluation of the Implementation of the Digital Transition Program A mixed methods approach will be used, combining quantitative and qualitative methods. Adolescents who participated in the digital program and healthcare providers will be included. The evaluation will focus on the intervention's reach, fidelity, perceived barriers, facilitators, usability, and user-friendliness of the digital platform.

TIMEPLAN The Digi-STEPSTONES project will be executed through six work packages, covering managerial, developmental, implementation, research, and reporting tasks, starting in 2023.

Ethical Approval The project has received ethical approval (2022-05394-01-351139, 2023-01-13).

By delivering the transition program digitally, Digi-STEPSTONES aims to reduce the burden on young patients, particularly those living in remote areas, and ensure that they receive the necessary transitional care. The project will contribute to Sweden's healthcare objectives by leveraging digital solutions to provide accessible, equitable, and high-quality care.

RESEARCH DESIGN AND METHODS

To address the specific objectives of this project, 2 studies will be conducted:

Objective 1 Study 1: Comparative effectiveness research: Non-inferiority trial Design: A two-arm, comparative, non-inferiority study, using a causal inference methodology will be performed. Arm A involves a pre-test/post-test design where individuals will participate in the digital delivery of the transition program.

Arm B is a historical comparison cohort that includes participants from two previous RCTs who received the intervention in-person.

Participants/inclusion criteria:

Arm A:

- Literate, Swedish-speaking adolescents with asthma/allergy or went through a solid organ transplantation aged minimum 15 years. Their parents will be invited to fill out a questionnaire (proxy).

Arm B:

* Literate, Swedish-speaking adolescents with asthma/allergy or went through a solid organ transplantation aged minimum 15 years. Their parents will be invited to fill out a questionnaire (proxy).

Sample size calculation:

Arm A: approximately 100 patients will be recruited consecutively Arm B: the approximate sample for individuals who received the intervention in-person is of approximately 120.

Exclusion criteria:

* Non literate
* Not Swedish speaking
* Cognitive impairment

Intervention: The STEPSTONES transition program is a multi-component intervention comprising 8 components: a) a transition coordinator (TC); b) information and education about the condition and treatment, health behavior, dealing with school and friends; c) availability by telephone; d) information about and contact with the adult program; e) guidance of parents; f) meeting with peers; g) person-centered transition plan; and h) the actual transfer to the adult program 15,16. These components are implemented in five steps: (1) first outpatient visit with TC; (2) second outpatient visit with TC; (3) information and peer-to-peer session for adolescents and their parents; (4) individualized transfer plan; and (5) actual transfer (Figure 2). The intervention will be delivered through the "Mitt vård mote" platform, which is currently being used across Sweden to undertake digital healthcare appointments. The HEADDDSS (home, education, activity, diet, drugs, depression, sex, safety) adolescent health interview is a cornerstone of the intervention. The intervention will be performed by specialized nurses of the respective pediatric care units, after being trained to become TC. The core of the STEPSTONES transition program remains the same for the present project, except that the delivery will be digital.

Variables and measurement: Assessments are planned at the age of 16 years (Time 0 - baseline ) and 18.5 years (Time 1- endpoint). The primary outcome is Patient Empowerment, using the Gothenburg Young Persons Empowerment Scale. Secondary outcomes are transition readiness; quality of life; and satisfaction with transition. In parents, the proxy transition readiness is measured.

Procedure of patient recruitment, data collection and data management: Patients who are eligible for inclusion will be approached by letter at the age of 16 years. In a subsequent telephone call, both the adolescents and their parents will be informed verbally about the study. Patients will only be included if the adolescent, who is a minor at the time of inclusion, provides written informed assent, and the parents/guardians provide written informed consent.

Patients will be asked to complete a set of online questionnaires (eCRF) online. To increase the response rate, a modified Dillman procedure will be used to minimize non-response, same procedure as in prior STEPSTONES trials. Reminders will be sent after three, five and seven weeks.

Statistical analysis: Propensity score weighting will be used as a method of causal inference. It mimics an RCT design and reduces comparative bias. After propensity weighting, the groups are compared by applying a linear model with doubly robust estimations. A one-sided p&amp;lt;0.025 will be used as the cutoff for statistical significance, because non-inferiority is hypothesized.

Objective 2 Study 2: Evaluation of the implementation of the digital transition program Design: for this evaluation, a mixed methods approach will be used, meaning a combination of quantitative and qualitative methods will be used.

Participants: adolescents who participated in the digital transition program as well as the nurses in charge of delivering the transition program (i.e., transition coordinators) will be included in this section. Additionally, personal from the adult healthcare unit will be interviewed.

Sample size: all participants from study 1 will be included in the quantitative assessment of this study. In the qualitative assessment, between 10-15 adolescents and around 10 healthcare providers will be interviewed.

Data collection: to describe the intervention's reach and fidelity, information on the number of participants that took part in the different components will be monitored. To identify perceived barriers and facilitators, as well as intervention fidelity, both the adolescents and healthcare providers will be interviewed individually. To evaluate the usability and user friendliness of the digital platform, a questionnaire will be answered. This questionnaire will be answered once they have finalized the transition program, meaning it will be included in the set of questionnaires the participants answer in study when they are 18,5 years. Lastly, a percentage of the digital meetings will be audio recorded and the care plans related to the intervention will be studied to understand the mechanism of delivery.

ELIGIBILITY:
Participants:

Arm A - Literate and Swedish-speaking adolescents with asthma/allergy or went through a solid organ transplantation aged minimum 15 years. Their parents will be asked to fill out one questionnaire (proxy).

Arm B:

- Literate and Swedish-speaking adolescents with asthma/allergy or went through a solid organ transplantation aged minimum 15 years. Their parents will be asked to fill out one questionnaire (proxy).

Sample size calculation:

Arm A: approximately100 patients will be recruited consecutively. Arm B: the approximate sample for individuals who received the intervention in-person is of

Ages: 15 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 100 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Patient empowerment | At baseline T0 when the participant is 16 years with follow up at T1 when the participants are 18.5 years
  Gothenburg Young Persons Empowerment Scale (GYPES)

SECONDARY OUTCOMES:
Satisfaction with transition | 18.5y
  Transitional care EXPeriences Questionnaire
Transition readiness | At baseline T0 when the participant is 16 years with follow up at T1 when the participants are 18.5 years
  Readiness for Transition Questionnaire (RTQ)- adolescent version

OTHER OUTCOMES:
Transition readiness | Parents fills out the questionnaire at baseline T0 when their adolescent (participant) is 16 years with follow up at T1 when the participant are 18.5 years
  Readiness for Transition Questionnaire (RTQ)-parent version PROXY

CONTACTS AND LOCATIONS:
Locations (2):
- Sweden (2):
  - Queen Silvia Childrens hospital, Sahlgrenska university hospital, Gothenburg, Vastra Gotalandsregionen
  - Institute of Health and Care Sciences, Sahlgrenska Academy, University of Gothenburg, Gothenburg

IPD SHARING:
Plan to Share IPD: Undecided
ethical considerations

REFERENCES:
- [Background] Vallmark M, Brorsson AL, Sparud-Lundin C, Bratt EL, Moons P, Saarijarvi M, Mora MA. Development and psychometric evaluation of TEXP-Q: a questionnaire measuring transition and transfer experiences in emerging adults with type 1 diabetes. J Patient Rep Outcomes. 2023 Nov 8;7(1):111. doi: 10.1186/s41687-023-00652-1. PMID 37938469
- [Background] Bratt EL, Mora MA, Sparud-Lundin C, Saarijarvi M, Burstrom A, Skogby S, Fernlund E, Fadl S, Rydberg A, Hanseus K, Kazamia K, Moons P. Effectiveness of the STEPSTONES Transition Program for Adolescents With Congenital Heart Disease-A Randomized Controlled Trial. J Adolesc Health. 2023 Oct;73(4):655-663. doi: 10.1016/j.jadohealth.2023.02.019. Epub 2023 Apr 8. PMID 37032211
- [Background] Saarijarvi M, Wallin L, Moons P, Gyllensten H, Bratt EL. Implementation fidelity of a transition program for adolescents with congenital heart disease: the STEPSTONES project. BMC Health Serv Res. 2022 Feb 5;22(1):153. doi: 10.1186/s12913-022-07549-7. PMID 35123454
- [Background] Saarijarvi M, Wallin L, Moons P, Gyllensten H, Bratt EL. Mechanisms of impact and experiences of a person-centred transition programme for adolescents with CHD: the Stepstones project. BMC Health Serv Res. 2021 Jun 10;21(1):573. doi: 10.1186/s12913-021-06567-1. PMID 34112174
- [Background] Brorsson AL, Bratt EL, Moons P, Ek A, Jelleryd E, Torbjornsdotter T, Sparud-Lundin C. Randomised controlled trial of a person-centred transition programme for adolescents with type 1 diabetes (STEPSTONES-DIAB): a study protocol. BMJ Open. 2020 Apr 14;10(4):e036496. doi: 10.1136/bmjopen-2019-036496. PMID 32295780
- [Background] Acuna Mora M, Saarijarvi M, Moons P, Sparud-Lundin C, Bratt EL, Goossens E. The Scope of Research on Transfer and Transition in Young Persons With Chronic Conditions. J Adolesc Health. 2019 Nov;65(5):581-589. doi: 10.1016/j.jadohealth.2019.07.014. Epub 2019 Sep 17. PMID 31540780
- [Background] Saarijarvi M, Wallin L, Moons P, Gyllensten H, Bratt EL. Transition program for adolescents with congenital heart disease in transition to adulthood: protocol for a mixed-method process evaluation study (the STEPSTONES project). BMJ Open. 2019 Aug 2;9(8):e028229. doi: 10.1136/bmjopen-2018-028229. PMID 31377699
- [Background] Acuna Mora M, Luyckx K, Sparud-Lundin C, Peeters M, van Staa A, Sattoe J, Bratt EL, Moons P. Patient empowerment in young persons with chronic conditions: Psychometric properties of the Gothenburg Young Persons Empowerment Scale (GYPES). PLoS One. 2018 Jul 20;13(7):e0201007. doi: 10.1371/journal.pone.0201007. eCollection 2018. PMID 30028863
- [Background] Acuna Mora M, Sparud-Lundin C, Bratt EL, Moons P. Person-centred transition programme to empower adolescents with congenital heart disease in the transition to adulthood: a study protocol for a hybrid randomised controlled trial (STEPSTONES project). BMJ Open. 2017 Apr 17;7(4):e014593. doi: 10.1136/bmjopen-2016-014593. PMID 28420661